CLINICAL TRIAL: NCT04147468
Title: Effectiveness of Functional Strength Training and Virtual Reality Games on Improving Arm Function in Children With Cerebral Palsy
Brief Title: Functional Strength Training and Virtual Reality in Children With CP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding has expired in June 2022. This protocol will be active once more funding is secured.
Sponsor: Georgia State University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Yuping Chen, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17349
Record Dates: First submitted 2019-10-08; First posted 2019-11-01 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: Virtual Reality; Functional Strength Training; Arm Function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: One group will receive virtual reality; the other group will receive functional strength training
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Gaming Intervention (Active Comparator): A newly developed VR gaming platform called Super Pop VR, a VR system that can be individualized to the movement capabilities of the child, will be used. The research team will loan the system to the family. The child will be asked to move their arms to 'pop' as many virtual objects as possible with the focus on outwards, upwards, and across midline.
  Interventions: Other: Virtual Reality
- Functional Strength Training (Experimental): Children will receive repetitive progressive resistance exercise during goal-directed functional activity with the children focus on the activity being performed. Children will be offered a pamphlet containing suggested functional arm exercises which are designed to move their arms.
  Interventions: Other: Functional Strength Training

INTERVENTIONS:
Other: Virtual Reality — For the VR intervention, we focus on using our developed VR gaming platform called Super Pop VR, a VR system that can be individualized to the movement capabilities of the participant. The research team will travel to the family to conduct the intervention to ensure the treatment adherence. The participants will be asked to move their arms to 'pop' as many virtual objects as possible.
  Arms: Virtual Reality Gaming Intervention
Other: Functional Strength Training — For the functional strength training, participants will receive repetitive progressive resistance exercise during goal-directed functional activity with the participants focus on the activity being performed. The research team will also go to the family to conduct the FST intervention.
  Arms: Functional Strength Training

SUMMARY:
Virtual reality (VR) has shown to be effective to improve arm function in children with cerebral palsy (CP). Recently, functional strength training (FST) starts to show to improve arm function in patients with stroke but has not been extensively explored in children with CP. This pilot study is to examine the effect of FST and VR on improving arm function in children with CP as well as the neuroplasticity changes in the brain related to the level of improvement.

Ten children with spastic CP will be recruited to participate in this pilot study. Children will be randomized to receive either VR of FST for 60 minutes per session x 3 sessions per week x 6 weeks at their home. All children will be evaluated prior to and immediately after the intervention at their home for clinical tests and at CABI for the MRI measures. Brain imaging data and clinical outcome measures including reaching kinematics, standardized fine motor assessment tool (Peabody Developmental Motor Scale-2nd edition), and daily use of affected hand (using Revised Pediatric Motor Activity Log) will be evaluated. A physical therapist who is blinded to the status will conduct the assessment.

The investigators anticipate children in both groups will improve their arm function after intervention; however, children in the VR group will have a better improvement as compared with children in the FST group.

ELIGIBILITY:
Inclusion Criteria:

* children with spastic CP are between ages 5-18 years; adults with spastic CP are between 19-30 years
* diagnosed with spastic CP
* have a Manual Ability Classification System (MACS) level I-III
* able to sit with trunk supported
* are able to reach forward for more than half of their arm length
* are able to follow three-step commands
* are able to see video screen (with or without corrected vision); and
* their primary caregiver is willing to follow the desired intervention "dosing" and all evaluation measurements, including MRI.

Exclusion Criteria:

* they have received surgery or botulinum toxin type A injection in the training arm within the preceding 4 months or are scheduled to receive it during the planned study period, or
* if they have a severe attention deficit or uncontrolled epilepsy which may possibly be triggered by the light or sound of the virtual reality games.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Brain neuroplasticity | Change from pre-intervention to the end of intervention, an average of 6 weeks
  Brain images of primary sensorimotor cortex (SMC), the premotor cortex (PMC), and the supplementary motor area (SMA). During MRI measures, fMRI will be used to investigate cortical activation during a rest condition and 3 task conditions: 1) visually-guided wrist movement, 2) passively-guided wrist movement, and 3) imagined wrist movement. The same visual display will be shown to the participants in all conditions.
Reaching kinematics | Change from pre-intervention to the end of intervention, an average of 6 weeks
  Reaching kinematics will be assessed while the child is interacting with Super Pop VRTM, wherein virtual bubbles are projected onto the TV in randomly dispersed locations, using the Kinect system. Three testing bubbles will be tested in the location where children need to reach about arm length overhead at 180, 135, and 90 degrees of shoulder abduction. Children's reaching kinematics will also be assessed while playing the real-life functional activity by inserting an envelope into a mailbox slip located in neutral, outward 45, and inward 45 using the Kinect system. Position data from the Kinect will be converted into 3-dimensional coordinate data and kinematic variables (movement time, trajectory straightness, speed, smoothness) will be computed.
Fine motor function | Change from pre-intervention to the end of intervention, an average of 6 weeks
  The fine motor domain of the Peabody Developmental Motor Scales, 2nd edition (PDMS-2) will be used. Two subsets of the Fine Motor Domain will be used to evaluate the children: grasping and visual-motor integration. Each item is rated as 0, 1, and 2 (0: child cannot attempt the item; 1: child's performance shows resemblance but not fully met the criteria; 2: child performs the item according to the criteria specified for mastery). Raw score will later be compared to the norm values and converted to percentile of the norm values.
Daily use of affected hand | Change from pre-intervention to the end of intervention, an average of 6 weeks
  Daily use of affected hand will be evaluated using Revised Pediatric Motor Activity Log (R-PMAL), which is filled out by primary caregivers about how often and how well their children use the affected arm in daily activities.

SECONDARY OUTCOMES:
Muscle strength | Change from pre-intervention to the end of intervention, an average of 6 weeks
  Muscle strength of shoulder flexion, extension, abductor, adduction, external rotation, and internal rotation, elbow flexion and extension, and wrist flexion and extension will be measured using hand-held dynamometer prior to and after intervention.
Spasticity | Change from pre-intervention to the end of intervention, an average of 6 weeks
  Spasticity of shoulder flexion, extension, abduction, adduction, external rotation, and internal rotation, elbow flexion and extension, and wrist flexion and extension will also be measured using the Modified Ashworth Scale. It contains a scale of 0 to 4 with 0 as no spasticity to 4 as rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Chen, ScD, PT, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No